CLINICAL TRIAL: NCT04116515
Title: The Narrative Effect of Active Video Games on Long-term Moderate-to-Vigorous Physical Activity (Main Trial)
Brief Title: Active Video Games on Physical Activity (Main Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Amy Lu, Associate Professor, Northeastern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK109316 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Physical Inactivity in Children
Keywords: Active Video Game; Physical Activity; Narrative; Child Obesity
MeSH Terms: conditions — Motor Activity; Narration; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be informed of their group at the conclusion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care Only (Active Comparator): A third of the participants will have standard clinical care only.
  Interventions: Behavioral: Standard clinical care
- Care + AVG (Experimental): A third of the participants will have the same standard clinical care plus an Xbox and active games.
  Interventions: Behavioral: Xbox / active video games; Behavioral: Standard clinical care
- Care + AVG + Narratives (Experimental): A third of the participants will have the same standard clinical care, an Xbox and active games, plus the stories delivered to their Xbox consoles.
  Interventions: Behavioral: Xbox / active video games; Behavioral: Animated cartoon narratives; Behavioral: Standard clinical care

INTERVENTIONS:
Behavioral: Xbox / active video games — The investigators would expect children to play active video games as a way to reduce their sedentary activities and increase their moderate and vigorous physical activities.
  Arms: Care + AVG; Care + AVG + Narratives
Behavioral: Animated cartoon narratives — The investigators would expect the animated cartoon narratives to motivate children to play more active video games as a way to reduce their sedentary activities and increase their moderate and vigorous physical activities.
  Arms: Care + AVG + Narratives
Behavioral: Standard clinical care — Each clinic will provide standard clinical care to the participants.

SUMMARY:
The purpose of the study is to test the effects of different versions of active video games (AVGs) on body composition, cardiometabolic risks, and cognitive functions among overweight/obese children over 6 months.

DETAILED DESCRIPTION:
The study aims to explore the effects of narrative-enhanced AVG on (1) body composition, (2) cardiometabolic risks, and (3) cognitive functioning among overweight/obese 8-12 years old children over 6 months.

A total of 210 children will be recruited from Tufts Floating Hospital, Boston Children's Hospital, and Martha Eliot Health Center. The investigators divided the participants into three groups to evaluate the effect of using active game consoles and stories to motivate children to exercise: A third of them have standard clinical care only; a third of them have the same standard clinical care plus an Xbox and active games; the remaining third of them have the same standard clinical care, an Xbox and active games, plus the stories delivered to their Xbox consoles.

Each child, accompanied by their guardian, will be asked to visit the Northeastern University Exercise Science Laboratory over the 6-month period. Blood samples, body composition (using Dual-energy X-ray absorptiometry, or DEXA Scan), and cognitive and affective evaluations of the active video games (AVGs) will be collected. Additionally, parents will be asked to fill out questionnaires related to their child's physical activity behaviors. Children would also be required to wear two accelerometers (essentially, a "smart watch" or activity tracker) on their wrist and waist for 7 consecutive days after the three visits within the 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 8-to-12-year-old
* Being overweight or obese (BMI% >=85)
* Speak and understand English
* Are willing and able to complete all measures
* Equal numbers of both genders will be recruited
* One child per household will be eligible to participate

Exclusion Criteria:

* Not between 8 and 12
* Not being overweight or obese
* Do not speak and understand English
* Have medical or physical problems that prevent them from playing AVGs, such as epilepsy
* Use orthopedic devices

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Changes in objective child physical activity | 6 months
  Physical activity will be measured with two 7-day accelerometer worn on the wrist and hip after three visits over 4-6 weeks, including minutes/day MVPA total. Physical activity and time spent in moderate to vigorous physical activity will be measured by two triaxial accelerometer (Actigraph Link and Actigraph GT3X+, Actigraph, Ft. Walton Beach, FL). Children will be asked to wear them for 7 full days during periods.
Changes in fat% | 6 months
  Measured through dual-energy X-ray absorptiometry (DEXA) scan by GE Lunar Prodigy (GE Healthcare, Chicago, IL).
Changes in lean tissue% | 6 months
  Measured through dual-energy X-ray absorptiometry (DEXA) scan by GE Lunar Prodigy (GE Healthcare, Chicago, IL).

SECONDARY OUTCOMES:
BMI% | 6 months
  The investigators plan to use the weight in kilograms and height in meters from the DEXA scan and children's birthdays and sex to calculate their BMI% using the CDC Calculator.
Fasting Insulin | 6 months
  Analysis of the plasma samples will be performed using dedicated Enzyme-Linked Immunosorbent Assay (ELISA) kits.
Fasting Glucose | 6 months
  Analysis of the plasma samples will be performed using dedicated Enzyme-Linked Immunosorbent Assay (ELISA) kits.
Lipid | 6 months
  Analysis of the serum samples will be performed using dedicated Enzyme-Linked Immunosorbent Assay (ELISA) kits.
C-reactive protein (CRP) | 6 months
  Analysis of the serum samples will be performed using dedicated Enzyme-Linked Immunosorbent Assay (ELISA) kits.

OTHER OUTCOMES:
Sustained Attention | 6 months
  Response time will be measured by the Psychomotor Vigilance Task
Working Memory | 6 months
  Response time will be measured by the Delayed Match-to-Sample Task
Working Memory | 6 months
  Response accuracy will be measured by the Delayed Match-to-Sample Task
Inhibitory Control | 6 months
  Response time will be measured by the Stroop Test
Inhibitory Control | 6 months
  Response accuracy will be measured by the Stroop Test
Physical Activity Motivation | 6 months
  Physical Activity Motivation will be measured by the Physical Activity Motivation scale through self-report

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lu AS, Baranowski T, Barreira TV, Fleischman A, Green MC, Huang SY, Lee IM, Levitsky LL, Noubary F, Thompson D. The impact of narratives and active video games among black and hispanic children with overweight and obesity: a randomized controlled trial. Int J Behav Nutr Phys Act. 2025 May 26;22(1):60. doi: 10.1186/s12966-025-01756-1. PMID 40420195